CLINICAL TRIAL: NCT04038515
Title: Impact of Flavors on Nicotine Perception and Self-Administration Via E-cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2000029704; R01DA046360 (NIH); 2000025408 (Other: Original IRB #)
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Nicotine; E-liquid Flavors
Keywords: Menthol; Electronic Nicotine Delivery Systems
MeSH Terms: conditions — Vaping | interventions — Nicotine; Menthol; Fruit

STUDY DESIGN:
Intervention Model Description: This is a within-subject, cross-over design. Participants will be invited to complete 4 test sessions. Across those 4 test sessions, participants will self-administer e-cigarettes containing all 20 e-liquid conditions (4 nicotine * 5 flavor conditions) in both 'directed' and ad libitum self-administration study components. The order of nicotine and flavor will be randomized across participants.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Although participants will receive all conditions in this within-subject cross-over study, the participant and researcher will be blinded to the order of e-liquid conditions (nicotine level, flavor) across and within test sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- E-liquid Order 'A' (Experimental): Order 'A' for E-liquid Self-Administration: All participants will be given all e-liquids (i.e., all 20 nicotine*flavor combinations (4 nicotine* 5 flavor combinations)) in this within-subject, cross-over design study. Participants will be randomized the order in which they self-administer the 20 nicotine*flavor combinations of e-liquid (across and within the 4 visits). The specific order cannot be described here without disrupting the double-blind nature of the study design.
  Interventions: Drug: Nicotine 0 mg/mL; Drug: Nicotine 6 mg/mL; Drug: Nicotine 12 mg/mL; Drug: Nicotine 24 mg/mL; Other: 'Menthol' flavor; Other: 'Menthol/Mint' flavor; Other: 'Green Apple' flavor; Other: 'Watermelon' flavor; Other: 'Unflavored'
- E-liquid Order 'B' (Experimental): Order 'B' for E-liquid Self-Administration: All participants will be given all e-liquids (i.e., all 20 nicotine*flavor combinations (4 nicotine* 5 flavor combinations)) in this within-subject, cross-over design study. Participants will be randomized the order in which they self-administer the 20 nicotine*flavor combinations of e-liquid (across and within the 4 visits). The specific order cannot be described here without disrupting the double-blind nature of the study design.
  Interventions: Drug: Nicotine 0 mg/mL; Drug: Nicotine 6 mg/mL; Drug: Nicotine 12 mg/mL; Drug: Nicotine 24 mg/mL; Other: 'Menthol' flavor; Other: 'Menthol/Mint' flavor; Other: 'Green Apple' flavor; Other: 'Watermelon' flavor; Other: 'Unflavored'
- E-liquid Order 'C' (Experimental): One nicotine level condition is a medium nicotine e-liquid (12 mg/mL nicotine). All participants will be given all e-liquids (i.e., all 20 nicotine*flavor combinations (4 nicotine* 5 flavor combinations)) in this within-subject, cross-over design study. Participants will be randomized the order in which they self-administer the 20 nicotine*flavor combinations of e-liquid (across and within the 4 visits). The specific order cannot be described here without disrupting the double-blind nature of the study design.
  Interventions: Drug: Nicotine 0 mg/mL; Drug: Nicotine 6 mg/mL; Drug: Nicotine 12 mg/mL; Drug: Nicotine 24 mg/mL; Other: 'Menthol' flavor; Other: 'Menthol/Mint' flavor; Other: 'Green Apple' flavor; Other: 'Watermelon' flavor; Other: 'Unflavored'
- E-liquid Order 'D' (Experimental): One nicotine level condition is a high nicotine e-liquid (24 mg/mL nicotine). All participants will be given all e-liquids (i.e., all 20 nicotine*flavor combinations (4 nicotine* 5 flavor combinations)) in this within-subject, cross-over design study. Participants will be randomized the order in which they self-administer the 20 nicotine*flavor combinations of e-liquid (across and within the 4 visits). The specific order cannot be described here without disrupting the double-blind nature of the study design.
  Interventions: Drug: Nicotine 0 mg/mL; Drug: Nicotine 6 mg/mL; Drug: Nicotine 12 mg/mL; Drug: Nicotine 24 mg/mL; Other: 'Menthol' flavor; Other: 'Menthol/Mint' flavor; Other: 'Green Apple' flavor; Other: 'Watermelon' flavor; Other: 'Unflavored'

INTERVENTIONS:
Drug: Nicotine 0 mg/mL — E-liquid containing no nicotine (0 mg/mL nicotine) will be self-administered via e-cigarettes. This will be administered in 5 flavor conditions (1 unflavored, 2 menthol, and 2 fruit conditions).
  Other Names: nicotine
Drug: Nicotine 6 mg/mL — E-liquid containing low nicotine (6 mg/mL nicotine) will be self-administered via e-cigarettes. This will be administered in 5 flavor conditions (1 unflavored, 2 menthol, and 2 fruit conditions).
  Other Names: nicotine
Drug: Nicotine 12 mg/mL — E-liquid containing medium nicotine ( 12 mg/mL nicotine) will be self-administered via e-cigarettes. This will be administered in 5 flavor conditions (1 unflavored, 2 menthol, and 2 fruit conditions).
  Other Names: nicotine
Drug: Nicotine 24 mg/mL — E-liquid containing high nicotine ( 24 mg/mL nicotine) will be self-administered via e-cigarettes. This will be administered in 5 flavor conditions (1 unflavored, 2 menthol, and 2 fruit conditions).
  Other Names: nicotine
Other: 'Menthol' flavor — E-liquid containing 'menthol' flavor will be self-administered via e-cigarettes. This will be administered in 4 nicotine conditions (0, 6, 12, 24 mg/mL nicotine).
  Other Names: menthol
Other: 'Menthol/Mint' flavor — E-liquid containing 'menthol/mint' flavor will be self-administered via e-cigarettes. This will be administered in 4 nicotine conditions (0, 6, 12, 24 mg/mL nicotine).
  Other Names: menthol
Other: 'Green Apple' flavor — E-liquid containing 'green apple' flavor will be self-administered via e-cigarettes. This will be administered in 4 nicotine conditions (0, 6, 12, 24 mg/mL nicotine).
  Other Names: fruit
Other: 'Watermelon' flavor — E-liquid containing 'watermelon' flavor will be self-administered via e-cigarettes. This will be administered in 4 nicotine conditions (0, 6, 12, 24 mg/mL nicotine).
  Other Names: fruit
Other: 'Unflavored' — E-liquid containing no additional flavor (i.e., 'unflavored') will be self-administered via e-cigarettes. This will be administered in 4 nicotine conditions (0, 6, 12, 24 mg/mL nicotine).
  Other Names: unflavored

SUMMARY:
The goal of this application is to test whether menthol and fruit flavors impact e-cigarette use through dissociable mechanisms and exert their effects differentially across nicotine doses.

DETAILED DESCRIPTION:
This study examines the impact of menthol and fruit flavors on self-administration of e-cigarette solutions containing varying amounts of nicotine. This is a randomized, double-blind study with a within-subject cross-over design, using e-liquids with 5 different flavors and 4 different levels of nicotine for a total of 20 different e-liquid formulations. Each subject will participate in 4 test sessions. The order of flavor and nicotine delivery will be randomized. At each test session, they will undergo directed self-administration, in a randomized order, then an ad libitum self-administration session where they can choose among all of the e-cigarettes used during the directed session. The primary aims assess the impacts of nicotine and flavor (and their interactions) on participants' subjective ratings of the e-liquids during the 'directed' self-administration component, and self-administered puffs during the ad libitum self-administration component. In addition, the study will explore the impact of sex/gender and sensitivity to nicotine aversiveness or bitterness (as operationalized by genetic variations in the alpha-5 subunit of nicotinic acetylcholine receptor that influences the aversive effects of nicotine, or a taste receptor number 38 ( TAS2R38) important for bitterness perception) on study outcomes.

ELIGIBILITY:
INCLUSION CRITERIA

* Aged 18 to 30;
* Past month daily nicotine-containing e-cigarette, cigarette, and/or cigar/little cigar/cigarillo use;
* Urine cotinine levels consistent with regular nicotine use (e.g., NicAlert urine cotinine dipstick ≥3 or Accutest Positive for Cotinine);
* For females, using acceptable birth control methods;
* Able to provide written informed consent;
* Able to read and write in English;
* Stated willingness to comply with all study procedures (including self-administration of all e-liquid conditions; attend in-person sessions; comply with COVID guidelines of the research facilities) and lifestyle considerations (including overnight nicotine abstinence) and availability for the duration of the study;
* Cardiovascular measures in normal/ non-hypertensive range for adults, including resting heart rate (HR) of 60-100 bpm; blood pressure (BP) of equal to or less than 129 mmHg (systolic)/80 mmHg (diastolic)); and oximeter (i.e., blood oxygenation) readings of 95-100 SpO2;
* Resident of the State of Connecticut.

Exclusion Criteria:

* Any allergy or known hypersensitivity to propylene glycol, vegetable glycerin, menthol, mint, green apple or watermelon flavorants or history of allergic or hypersensitive reaction to use of an e-cigarette/vaping device;
* Has not used e-cigarettes at least 10 times in the last 6 months;
* For females, pregnant (as determined by pregnancy screening) or breast feeding;
* Seeking (or undergoing) treatment for nicotine dependence or tobacco product use (smoking or vaping) or has current plans to quit tobacco product use;
* Meet current criteria for psychiatric disorder (according to the MINI);
* Current or history of respiratory illnesses including pneumonia with COVID-19 , other medical illness, and/or psychotropic medication use that a clinician investigator deems a contraindication for study participation.
* History of environmental - bronchospastic allergies, multiple chemical sensitivities, or other airway sensitivities that require the use of an epi pen or that in the investigators view would make it risky for participation;
* Not fully vaccinated for COVID-19

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Subjective drug ratings | immediately after intervention
  Subjective ratings of e-liquids delivered via e-cigarette will be assessed during the 'directed' self-administration component of each test day, using visual analogue scales (VAS). VAS scores range from 0=not at all to 100=extremely. Separate VAS scales will be collected for subjective ratings of aversive properties (higher scores reflect more aversiveness) and rewarding properties (higher scores reflect more rewarding properties) of the e-cigarettes, in each nicotine*flavor condition. Subjective drug ratings for each nicotine*flavor condition will be tested at one test day only and the order of nicotine*flavor conditions will be randomized across the test days (and order within test days will be randomized).
E-cigarette use | immediately after intervention
  Number of puffs from each e-cigarette (containing different e-liquids) will be measured during the ad libitum self-administration component of each test day. E-cigarette use (ad libitum puffs) for each nicotine*flavor condition will be tested at one test day only and the order of nicotine*flavor conditions will be randomized across the test days (and order within test days will be randomized).

CONTACTS AND LOCATIONS:
Overall Officials: Elise DeVito, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No